CLINICAL TRIAL: NCT01624597
Title: A Randomized Controlled Trial to Improve Teen Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Corinne Peek-Asa, Professor, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 065095; R01HD065095 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Motor Vehicle Driving
Keywords: Road traffic safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Participants will have a passive in-vehicle video device installed in their car to measure driving errors and safety behaviors.
- In-vehicle video feedback (Experimental): Participants will receive feedback from an in-vehicle video system. A light on the system will blink when a driving event has been recorded. Parents will receive a weekly report card of driving errors.
  Interventions: Behavioral: In-vehicle video feedback; Behavioral: Parent communication
- In-vehicle video feedback, parent communication (Experimental): Participants will receive feedback from an in-vehicle video system. A light on the system will blink when a driving event has been recorded. Parents will receive a weekly report card of driving errors. Parents will participate in an intervention that provides input on teaching and communicating about driving skills and safety behaviors.
  Interventions: Behavioral: Parent communication

INTERVENTIONS:
Behavioral: In-vehicle video feedback — An in-vehicle video system will record driving errors and safety behaviors. A light on the system will blink to let the participant know that a driving error has been recorded. Parents will receive a weekly report card.
  Arms: In-vehicle video feedback
Behavioral: Parent communication — Parents will receive instruction in teaching and effective communication about driving skills and driving safety. The intervention includes driving goals for teen drivers and parent communication strategies.
  Arms: In-vehicle video feedback; In-vehicle video feedback, parent communication

SUMMARY:
This randomized controlled trial will evaluate an intervention that provides parents with objective feedback about their teen's driving as well as strategies to improve communication with their teen about driving. We will recruit 180 newly-licensed teen drivers and a parent or guardian. Our main hypotheses are that: parent-teen dyads who receive feedback will have reduced driving errors and increased safety behaviors than dyads with no feedback; and, parent-teen dyads who receive instruction on communication techniques will have improved quality and quantity of communication about driving than dyads not learning these techniques.

DETAILED DESCRIPTION:
With a long-range goal of reducing crashes and related injuries among teen drivers, this project will assess the influence of a parent-focused intervention on teens' driving and safety behaviors. This randomized controlled trial will evaluate an intervention that integrates an in-vehicle video feedback system with parent-based communication techniques to improve teen driving. This will be the first rigorous evaluation of this technology, as well as the first to integrate a parent component. The in-vehicle video system records a video clip whenever an abrupt change in speed or steering direction is detected. These event-triggered video clips will be coded to identify safety-relevant events like driving errors and safety behaviors. A randomized group of parents will receive a weekly "driving report card" that summarizes driving errors, safety behaviors, and crashes or near-crashes recorded by the in-vehicle system. A second group of randomized parents will receive the report card plus training in communication strategies specifically designed to improve parent-teen communication about safe driving (based on Motivational Interviewing). Driving errors and safety behaviors will be compared to a control group that receives no feedback from the in-vehicle video system.

The specific aims of this proposed project are:

Specific Aim 1: Identify if giving parents feedback about their teen's driving performance and skills to better communicate with their teen driver increases the quality and quantity of parental involvement in teen driving.

Hypothesis: The intervention groups will report more frequent and higher-quality communication about safe driving than the control group.

Specific Aim 2: Identify if giving parents feedback about their teen's driving performance and skills to better communicate with their teen driver decreases the frequency of driving errors, unsafe driving behaviors, crashes, and near crashes.

Hypothesis: The intervention groups will have significantly reduced risky driving events (driving errors, crashes, and near crashes) and significantly increased safety behaviors (such as safety belt use and driving without distractions) than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Teen will receive Intermediate Driver's license in three months
* Teen has regular access to a car
* Can provide proof of insurance
* One legal guardian will also consent to participation

Exclusion Criteria:

* Either parent or teen is not an English speaker
* A sibling has already participated in the study

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Driving errors by newly licensed teen drivers | 6 months after licensure
  An in-vehicle video system will be used to measure driving errors made by newly licensed teen drivers

SECONDARY OUTCOMES:
Safety behaviors of newly licensed teen drivers | 6 months post-licensure
  An in-vehicle video system will be used to measure safety behaviors practiced by newly licensed teen drivers.
Parent communication | 6 months
  Parents and teens will report on communication quality and quantity related to safe driving.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Peek-Asa, PhD, Principal Investigator — University of Iowa; Daniel McGehee, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa